CLINICAL TRIAL: NCT01286324
Title: A Pilot Grant to Examine the Feasibility, Efficacy and Tolerability of a Standardized Chamomile Extract in Treating Chronic Primary Insomnia
Brief Title: Chamomile for Chronic Primary Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Suzanna Zick, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101,749
Record Dates: First submitted 2011-01-24; First posted 2011-01-31 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Primary Insomnia; Chronic Insomnia
Keywords: Matricaria; Chamomile; Herb; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chamomile High Grade Extract (Experimental): Each capsule contains 90 mg dry extract of chamomile flowering tops [6:1 (v/v) extraction solvent (ethanol 70%/30% water): flowering tops] standardized up to 2.5 mg of (-)-α-bisabolol and ≥ 2.5 mg of apigenin per tablet
  Interventions: Dietary Supplement: Chamomile High Grade Extract
- Placebo Tablet (Placebo Comparator): Contained lactose
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Dietary Supplement: Chamomile High Grade Extract — three tablets each (equivalent to 7.5 g of dried herb) p.o. twice daily for 28 days
  Arms: Chamomile High Grade Extract
Drug: Placebo Tablet
  Arms: Placebo Tablet

SUMMARY:
The purpose of this study is to determine if an herb called chamomile can help to treat insomnia (difficulty in going to sleep or getting enough sleep) by increasing the amount of time that you sleep and/or improving the quality of your sleep. The study will also be looking at the effect of chamomile on day time fatigue and functioning.

DETAILED DESCRIPTION:
Insomnia, defined as the inability to initiate or maintain sleep or lack of restorative sleep, is the most prevalent sleep complaint in primary care. Insomnia is associated with decreased quality of life, work limitations and increased healthcare utilization. Currently there is no treatment for chronic insomnia that is readily available, affordable, without significant side-effects and demonstrated to be safe for long term use. Consequently, treatments that would fill this gap are needed.

Chamomile (Matricaria recutita) has been used as a gentle sleep agent by herbalists for several hundred years. It has been studied in animals for its sedative potential and shows promise for treating insomnia. Currently, chamomile's sedative mechanisms of action are unknown, but are thought to be through the major inhibitory neurotransmitter in the central nervous system, γ - aminobutyric acid (GABA). However, no study has examined chamomile's efficacy and safety for treating insomnia.

The investigators propose a double-blind, placebo-controlled, randomized trial of chamomile in primary care patients with chronic insomnia. Thirty-four patients will be randomized to either Chamomile High Grade Extract, three 5 mg tablets standardized to 0.4% (-)-α-bisabolol twice daily or placebo and will be followed for 28 days for changes in a sleep diary (sleep efficiency, total sleep time, sleep-onset latency and sleep quality), insomnia severity and sleep disturbances. Secondary endpoints include assessing changes in day time functioning (measures of global quality of life, depression and anxiety) and monitoring for any signs of toxicity. The investigators will also determine the feasibility of conducting a larger trial with this agent.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 64 years;
* Must be able to give written informed consent;
* Have a diagnosis of primary insomnia per DSM-IV criteria, reporting < 6.5 hours sleep and/or >30 minutes to fall asleep (SOL) and/or wake after sleep onset (WASO) > 30 minutes, three or more nights per week;
* Present sleep complaint for at least 6 months;

Exclusion Criteria:

* Women who are pregnant, lactating or less than six months post-partum. Due to the fact that an assessment of reproductive performance and teratology tests have not been conducted we are excluding pregnant and lactating women;
* Patients with unstable medical conditions;
* DSM-IV Axis I or personality disorder diagnosis with the exception of patients with treated and stable unipolar depression or generalized anxiety disorder (such that the PRIME-MD scores are within normal range for these disorders);
* Difficulty in sleep initiation or maintenance associated with known medical diagnosis or conditions that may affect sleep, e.g., sleep apnea, restless leg syndrome, chronic pain;
* Evidence of lack of reliability or noncompliance as defined by missing a pretreatment appointment more than twice;
* Current diagnosis of substance abuse or dependence;
* Known allergy to chamomile or members of the ragweed family;
* Currently taking cyclosporine, warfarin or chronic sedative and anxiolytic medications;
* Prior use of insomnia medications is not exclusionary, but patients must be off of these medications at the screening visit and through out the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna M Zick, ND, MPH, Principal Investigator — University of Michigan; J. Todd Arnedt, PhD, Study Director — University of Michigan
Locations (1):
- University of Michigan Department of Family Medicine, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Zick SM, Wright BD, Sen A, Arnedt JT. Preliminary examination of the efficacy and safety of a standardized chamomile extract for chronic primary insomnia: a randomized placebo-controlled pilot study. BMC Complement Altern Med. 2011 Sep 22;11:78. doi: 10.1186/1472-6882-11-78. PMID 21939549

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Tablet | Chamomile High Grade Extract
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Tablet | Chamomile High Grade Extract | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (15.3) | 42.2 (13.5) | 41.4 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Chamomile Extract on Measures of Sleep at Day 28.
Description: Change from baseline of chamomile extract, three tablets (equivalent to 7.5 g of dried herb) p.o. twice times daily versus placebo on the following sleep measures at 28 days:
  * the change from baseline of daily self-report of sleep as assessed by a sleep diary that includes determination of: (i) sleep efficiency, which equals "The total sleep time divided by time-in-bed, multiplied by 100." This measure is our primary aim (SE).
Time Frame: baseline and day 28
Measure: Least Squares Mean (Standard Deviation); unit: percentage of time asleep
Arm/Group | Placebo Tablet | Chamomile High Grade Extract
Number analyzed (Participants) | 17 | 17
percentage of time asleep | 83.3 (7.7) | 77.5 (12.9)
Statistical Analysis 1: Comparison: Placebo Tablet vs Chamomile High Grade Extract; Test type: Superiority; p = 0.21, t-test, 2 sided — Adjusted p-value based on a general linear model adjusted for group and the baseline of the measure

2. Secondary Outcome: Change From Baseline of Chamomile on Daytime Functioning Measures: BDI
Description: Change from baseline of chamomile extract, three tablets p.o. twice times daily versus placebo on daytime functioning measures at 28 days:
  * the change from baseline of measures of depression and anxiety evaluated respectively with the Beck Depression Inventory-II (BDI-II), which is scored on a scale of 0 to 63 where a total score of 0-13 is considered minimal range (minimal depression), 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: baseline and day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Tablet | Chamomile High Grade Extract
Number analyzed (Participants) | 17 | 17
units on a scale
  Pre-treatment | 6.0 (6.0) | 3.2 (1.6)
  Post-treatment | 4.8 (5.0) | 2.4 (2.4)
Statistical Analysis 1: Comparison: Placebo Tablet vs Chamomile High Grade Extract; Test type: Superiority; p = 0.60, t-test, 2 sided — Adjusted p-value based on a general linear model adjusted for group and the baseline of the measure

3. Secondary Outcome: Change From Baseline of Chamomile on Daytime Functioning Measures: STAI
Description: Change From Baseline of Chamomile on Daytime Functioning Measures, depression and anxiety evaluated respectively with the Beck Depression Inventory-II (BDI-II) and trait portrait of the State Trait Anxiety Index (STAI). STAI scores range for each subtest from 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the S-Anxiety scale
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Tablet | Chamomile High Grade Extract
Number analyzed (Participants) | 17 | 17
units on a scale
  Pre-Treatment State Subscale | 33.2 (9.7) | 30.8 (8.0)
  Post-treatment State Subscale | 33.6 (11.0) | 30.1 (6.8)
  Pre-Treatment Trait Subscale | 37.5 (11.3) | 36.3 (10.1)
  Post-Treatment Trait Subscale | 40.8 (15.5) | 35.5 (11.0)
Statistical Analysis 1: Comparison: Placebo Tablet vs Chamomile High Grade Extract; Statistical Analysis for State Subscale; Test type: Superiority; p = 0.47, t-test, 2 sided — Adjusted p-value based on a general linear model adjusted for group and the baseline of the measure
Statistical Analysis 2: Comparison: Placebo Tablet vs Chamomile High Grade Extract; P-value for Trait Subscale; Test type: Superiority; p = 0.45, t-test, 2 sided — Adjusted p-value based on a general linear model adjusted for group and the baseline of the measure

4. Secondary Outcome: Change From Baseline of Chamomile on Daytime Functioning Measures: Fatigue Severity Scale
Description: Change From Baseline of Chamomile on Daytime Functioning Measures: Fatigue Severity Scale (FSS) Range: 9 to 63. The 9-item scale measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders.
  The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Tablet | Chamomile High Grade Extract
Number analyzed (Participants) | 17 | 17
units on a scale
  Pre-Treatment FSS score | 30.9 (9.1) | 32.1 (10.6)
  Post-treatment FSS score | 32.3 (10.0) | 27.9 (9.3)
Statistical Analysis 1: Comparison: Placebo Tablet vs Chamomile High Grade Extract; Test type: Superiority; p = 0.11, t-test, 2 sided — P value is adjusted based on a general linear model adjusted for group and the baseline of the measure

5. Secondary Outcome: Change From Baseline of Chamomile on Daytime Functioning Measures [ Time Frame: Baseline and Day 28 ]
Description: the change from baseline of global QOL (as determined by the 12 Item Short Form Health Survey Version 2 {SF-12 V2})
Time Frame: Baseline and 28 days
Population: Before first participants completed the study, the decision was made not to gather this data for reasons of cost.
Arm/Group | Placebo Tablet | Chamomile High Grade Extract
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Changes From Baseline in the Safety and Tolerability of Chamomile
Description: Changes from baseline in the safety and tolerability of Chamomile High Grade Extract, three tablets (equivalent to 7.5g of dried herb) p.o. twice times daily versus placebo were measured by counting all participants who reported a serious or non-serious adverse event at the weekly check-ins that were established.
Time Frame: once per week during study and day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Tablet | Chamomile High Grade Extract
Number analyzed (Participants) | 17 | 17
Participants | 10 | 6

ADVERSE EVENTS:
Arm/Group | Placebo Tablet | Chamomile High Grade Extract
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 10/17 | 6/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Tablet (N=17) | Chamomile High Grade Extract (N=17)
Infections (Infections and infestations) | 3 | 2
Headaches (General disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
GI Symptoms (Gastrointestinal disorders) | 4 | 2
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
Used subjective sleep measures. We did not assess the characteristics of participants' sleep difficulties and these sleep issues may be important considering the age-range of individuals included in the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes